CLINICAL TRIAL: NCT03705650
Title: SHAPE: Seeing the Heart With AI Powered Echo
Brief Title: SHAPE:SeeingtheHeartwithAIPoweredEcho
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Guttas (Industry)
Responsible Party: Sponsor-Investigator, Sara Guttas, Clinical Applications Manager at Bay Labs, Caption Health, Inc.
Organization: Caption Health, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHAPE01
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Disease
Keywords: Disease detection; Medicare aged patients; routine physical examination; primary care; limited echocardiogram
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Medicare Primary Care Provider (PCP) Patients (Experimental): This is a non-randomized study of non-significant risk (NSR) that will be conducted at Northwestern's Central Dupage Hospital. Medicare patients > 65 years who are scheduled for a routine physical exam with their PCP that meet inclusion and exclusion criteria will be asked to participate in this study. Consenting patients will be scheduled for 2 back to back ultrasound scans including 5 standard 2D echocardiogram views each. The first scan will be performed by a non-ultrasound specialist using EchoGPS experimental guidance technology and the second control exam will be performed by a trained sonographer using a cleared conventional ultrasound platform.
  Interventions: Diagnostic Test: Limited Echocardiogram

INTERVENTIONS:
Diagnostic Test: Limited Echocardiogram — STUDY SOFTWARE non-significant risk (NSR) Bay Labs EchoGPS software interfaced with the Terason uSmart 3200t FDA 510(k)-cleared, commercially available ultrasound EchoGPS software communicates with the ultrasound image formation engine of the 510(k)-cleared Terason uSmart 3200t through an application programming interface (API). EchoGPS will be used to provide visual guidance, feedback and interpretation assistance to users during image acquisition. For this study, CMAs will use EchoGPS to perform point-of-care echocardiogram examinations.

SUMMARY:
Establish transthoracic echocardiogram (TTE) exams performed with Bay Labs EchoGPS guidance technology can be used in a primary care setting to accurately identify cardiac disease. In Phase I TTE exams with EchoGPS will be compared to findings from a commercially available, FDA 510(k)-cleared reference device (Terason uSmart 3200t, point-of-care ultrasound) without EchoGPS assistance technology. Study is non-significant risk (NSR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for a standard physical examination
2. Patients ≥65 years old

For patients in Phase I, one of the following additional inclusion criteria must be present:

1. Patient presenting with a new murmur, or history of a murmur but no prior echo within 3 years of the exam
2. Patient presenting with shortness of breath
3. Unexplained pedal edema

Exclusion Criteria:

1. Unable to lie flat for study
2. Significant anatomical abnormality, recent trauma, or recent thoracic/abdominal surgery that would limit the ability to obtain adequate images
3. Subjects unwilling or unable to give written informed consent
4. Patients experiencing a known or suspected acute cardiac event Eligibility criteria for Phases II and III of this study will be finalized once results from Phase I are available. The current plan is to have similar criteria for Phases II and III.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
% of diagnostic quality clips acquired by a non-specialist using experimental guidance software, with quality assessed using the American College of Emergency Physician (ACEP) Suggested Quality Assurance Grading Scale | 1 year
  All of the echo views (or "clips") acquired by non-specialists during the study will be scored for image quality (IQ) by clinicians using the 1-5 ACEP quality grading scale. In this scale, a score of 1 represents the poorest IQ and 5 the highest. Images must have a score of 3 or higher to be considered diagnostic quality. Diagnostic quality images (3+) meet at least minimal criteria for diagnosis to be supported and are therefore clinically acceptable.

SECONDARY OUTCOMES:
Number of minutes for non-specialists to perform studies using EchoGPS experimental guidance software | 1 year
  Number of minutes for non-specialists to perform studies using EchoGPS software as compared to that of the time for expert sonographer's control studies using FDA 510(k)-cleared, commercially available ultrasound platform. The time of Study Exam will be compared to that of Control Exam on a per subject basis (paired difference) for Phase I of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial, Central DuPage, Winfield, Illinois, United States